CLINICAL TRIAL: NCT05658198
Title: A Non-controlled Trial to Determine Whether Counseling Around HPV Increases Vaccine Uptake in Unvaccinated Patients Ages 18-35 Visiting a Rural Health Clinic for Primary or Reproductive Health-related Care in the Mississippi Delta
Brief Title: Investigating HPV Vaccination Uptake in Adults Aged 18-35 Seeking Care at a Health Clinic in Rural Mississippi
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Plan A Health, Inc (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 02
Record Dates: First submitted 2022-12-09; First posted 2022-12-20 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Human Papillomavirus Vaccination
Keywords: HPV vaccine; Gardasil; unvaccinated; adults
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Unvaccinated patients: Patients who are unvaccinated against HPV when they arrive at Plan A.
  Interventions: Behavioral: Counseling

INTERVENTIONS:
Behavioral: Counseling — Patients who first decline HPV vaccination receive a 3-5 minute counseling session on HPV and the benefits of the vaccine.

SUMMARY:
A study evaluating HPV vaccine uptake among unvaccinated patients between the ages of 18 and 35 of a mobile health clinic serving the Mississippi Delta.

DETAILED DESCRIPTION:
This study is intended to serve several purposes. The first is to determine whether patients between the ages of 18 and 35 visiting a mobile health clinic or brick and mortar clinic in the Mississippi Delta who have not received the HPV vaccine or have not completed the vaccine series are receptive to receiving it while seeking care. The second purpose is to determine whether those patients who initially decline the HPV vaccine are interested in receiving it after being counseled about HPV and the potential effects of the virus. The third purpose is to assess whether there is a statistically significant difference between the type of visit people who opt to receive the vaccine are making to the clinics. Finally, the knowledge, attitudes, and perceptions around HPV and the HPV vaccine will be assessed via group interviews with eligible participants at the conclusion of the study.

The study also includes two secondary objectives. The first is to assess whether adults who are not vaccinated against HPV are interested in receiving it. The second is to assess whether adults accurately recall whether they received a specific vaccine during childhood. The implications from these two objectives have the potential to influence policy changes regarding vaccine catch-up among adults and health communication practices as young adults transition out of pediatric care.

Anyone between the ages of 18 and 35 whose vaccination status can be verified is eligible to be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 and 35 and have a verified vaccine record that shows they were not vaccinated with the HPV vaccine or have not had a complete series of the vaccine before their visit.

Exclusion Criteria:

* patients who have been vaccinated against HPV
* patients under 18 and over 35
* patients whose vaccine records cannot be verified

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients between the ages of 18 and 35 visiting a primarily mobile health clinic in the Mississippi Delta.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Increased HPV vaccination rates | one year
  Determine whether offering the HPV vaccine free of charge to unvaccinated adults aged 18-35 receiving SRH or primary care services at a primarily mobile health clinic serving mainly low-income patients of color changes vaccination rates in the community.
Counseling effectiveness | one year
  Determine whether a 3-5 minute education session on HPV and HPV-related diseases for people who decline initial vaccination changes their vaccination intentions.
Visit differences | one year
  Determine whether a significant difference exists between the type of visit (SRH versus primary care) patients who decide to become vaccinated made to the clinic.
Prior information | one year
  Examine how access to and prior information given on the HPV vaccine, as well as risk assessment for HPV infection versus vaccination, among unvaccinated adults between 18 and 35, addresses vaccine discordancy and affects the decision to become vaccinated as an adult.

SECONDARY OUTCOMES:
Vaccine interest | one year
  To identify whether adults who are not vaccinated against HPV are interested in receiving the vaccine.

CONTACTS AND LOCATIONS:
Locations (1):
- Plan A Health, Inc, Louise, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] United Health Foundation, America's Health Rankings Annual Report. Accessed 15 March, 2022 at: https://www.americashealthrankings.org/explore/annual/measure/Immunize_HPV/state/ALL
- [Background] Mississippi State Department of Health (2018). Mississippi State Plan for Comprehensive Cancer Control 2018-2022. Retrieved 25 April, 2022.
- [Background] United States Census Bureau (2022). Health Insurance Coverage Status by Sex and Age, Mississippi. Retrieved 25 April, 2022.
- [Background] Meites E, Szilagyi PG, Chesson HW, Unger ER, Romero JR, Markowitz LE. Human Papillomavirus Vaccination for Adults: Updated Recommendations of the Advisory Committee on Immunization Practices. MMWR Morb Mortal Wkly Rep. 2019 Aug 16;68(32):698-702. doi: 10.15585/mmwr.mm6832a3. PMID 31415491
- [Background] Fowler, C. I., Gable, J., & Lasater, B. (2021, September). Family Planning Annual Report: 2020 National Summary. Washington, DC: Office of Population Affairs, Office of the Assistant Secretary for Health, Department of Health and Human Services.
- [Background] Cates JR, Brewer NT, Fazekas KI, Mitchell CE, Smith JS. Racial differences in HPV knowledge, HPV vaccine acceptability, and related beliefs among rural, southern women. J Rural Health. 2009 Winter;25(1):93-7. doi: 10.1111/j.1748-0361.2009.00204.x. PMID 19166567
- [Background] Hamborsky, J., & Kroger, A. (Eds.). (2015). Epidemiology and prevention of vaccine-preventable diseases, E-Book: The Pink Book. Public Health Foundation.
- [Background] Christy K, Kandasamy S, Majid U, Farrah K, Vanstone M. Understanding Black Women's Perspectives and Experiences of Cervical Cancer Screening: A Systematic Review and Qualitative Meta-synthesis. J Health Care Poor Underserved. 2021;32(4):1675-1697. doi: 10.1353/hpu.2021.0159. PMID 34803036